CLINICAL TRIAL: NCT03443037
Title: Benefits of Amantadine in Patients With Coma State
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Begum Ergan, Staff in the department of pulmonary and critical care medicine, Dokuz Eylul University
Other Study IDs: 265-SBKAEK
Record Dates: First submitted 2018-02-16; First posted 2018-02-22 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Coma; Prolonged; Amantadine
Keywords: Coma; Disability; amantadine
MeSH Terms: conditions — Coma | interventions — Amantadine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Amantadine group: Patients admitted to the critical care with diagnosis of coma state who have received amantadin 200 mg / day for fourteen days according to İCU protocols decided by primary physician
  Interventions: Drug: amantadine sulphate
- Control group: Patients admitted to the critical care with diagnosis of coma state who haven't received amantadin

INTERVENTIONS:
Drug: amantadine sulphate
  Groups: Amantadine group

SUMMARY:
The study was a single center observational-prospective study and approved by local ethics committee. Patients in coma state due to traumatic brain injury, cardiac arrest or ischemic stroke who are older than 18 years of age were included in the study. Patients who received amantadine 200mg/day for fourteen days according to ICU protocols decided by primary physician formed the amantadine group, and the rest of the subjects were included in the control group. All patients were evaluated for Glasgow Coma Score, JFK Coma Recovery Scale and Disability Rating Scale once a week for three months.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years, ≤ 65 years
* GCS score ≤ 8
* Coma state due to ischemic stroke, brain hemorhage, anoxic brain damage

Exclusion Criteria:

* <18 years, > 65 years
* Patients admitted to the critical care without diagnosis of coma state
* Patients admitted to critical care with coma state that are not duo to ischemic stroke, brain hemorhage, anoxic brain damage
* Metastatic malignant neoplazm
* Congenital or acquired brain function problem (cerebral palsy, autism etc)
* Patients with amantadine allergy
* Progressive degenerative diseases (Alzheimer, Parkinson diseases etc)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the coma state duo to ischemic stroke, brain hemorhage, anoxic brain damage included in this study.
Sampling Method: Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2016-03-01 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Glascow Coma Score | 1. At the time of enrollment 2. 12 weeks after the enrollment
  Glascow Coma Score

CONTACTS AND LOCATIONS:
Overall Officials: Necati Gokmen, MD, Study Chair — Dokuz Eylul University; Kutlay Aydin, Principal Investigator — Dokuz Eylul University; Kutlay Aydin, Study Director — Dokuz Eylul University; Begum Ergan, Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No